CLINICAL TRIAL: NCT06641791
Title: A Phase III Randomized Controlled Trial Comparing Palliative Stereotactic Body Radiotherapy vs. Palliative Standard Radiotherapy in Patients With Advanced Head and Neck Cancer
Brief Title: Palliative Steroeotactic Body Radiotherapy vs Palliative Standard Radiotherapy in Patients With Advanced Head and Neck Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN13
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Advanced Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Radiotherapy (SRT) (Active Comparator)
  Interventions: Radiation: Standard Radiotherapy (SRT)
- Stereotactic Body Radioterapy (SBRT) (Experimental)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Standard Radiotherapy (SRT) — 2400 cGy in 3 fractions - day 0/7/21, OR, 2500 cGy in 5 fractions over 1 week
  Arms: Standard Radiotherapy (SRT)
Radiation: Stereotactic Body Radiotherapy (SBRT) — 4500 cGy in 5 fractions (twice a week to primary and nodal GTV, OR, 4000 cGy in 5 fractions twice a week if organs at risk.
  Arms: Stereotactic Body Radioterapy (SBRT)

SUMMARY:
This study is being done to answer the following question: Does stereotactic body radiation therapy (SBRT) provide better cancer control compared to standard radiation therapy (RT) for those with advanced head and neck cancer?

DETAILED DESCRIPTION:
Stereotactic body radiation therapy, or SBRT, is a cancer treatment that more precisely delivers radiation to the tumour area with less radiation going to unaffected areas around the tumour. It uses fewer treatments of higher doses compared to standard radiation therapy.

This study is being done to find out if this approach is better than the usual approach for advanced head and neck cancer. The usual approach is defined as care most people get for advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mucosal squamous cell carcinoma (SCC) of the head and neck arising from at least one of the following sites: oro/hypopharynx, oral cavity, supraglottic larynx, maxillary sinus, nasal cavity, or unknown primary
* Stages TX or T0-T4/N0-N3
* Must be considered unfit for curative intent RT as determined by the treating oncologist(s)
* Geriatric 8 score <14
* Patient must be ≥18 years of age
* Staging CT or MRI of the head and neck within 8 weeks prior to randomization
* Chest CT or x-ray. PET CT is permitted if CT is of diagnostic quality.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-3
* Participants of childbearing potential must have agreed to use a highly effective contraceptive method during protocol therapy.
* Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational treatment are eligible for this trial.

Exclusion Criteria:

* Patients with nasopharyngeal carcinoma.
* Prior systemic therapy (including immunotherapy).
* Prior radiotherapy to the head and neck excluding superficial radiotherapy for head and neck skin cancer that does not overlap with current protocol treatment.
* Prior head and neck cancer excluding skin cancer.
* Patients with tumour locations/at risk of SBRT toxicity, including glottic/subglottic larynx, T4 hypopharynx, post-cricoid, cervical esophagus, circumferential pharyngeal involvement, extension/proximity to brain/optic structures, any single tumour mass >8 cm (in one dimension).
* > 2 nodal levels (Level 1a/b not counted); retropharyngeal lymph nodes (where the closest edge is < 2cm from the closest edge of CTV (primary or nodal) will not be considered as a different level). Note: a single lymph node mass that spans 2 levels will be considered as 1 level.
* Gross tumour poorly visualized on CT/MRI.
* Definitive radiological or clinically evident distant metastases.
* Scleroderma/CREST syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival estimated according to Kaplan-Meier's methodology | 6 years

SECONDARY OUTCOMES:
Progression-free Survival | 6 years
Local Regional Failure Free Survival | 6 years
  defined as the time from the date of randomization to the date of any of the following, whichever comes first:
  * The first record of appearance (radiological or clinical) of local or regional disease progression/recurrence.
  * Surgery of primary tumour at any time performed for clinical or radiological (RECIST 1.1) disease persistence/progression/recurrence with tumour present/unknown on final pathology.
  * Neck dissection > 20 weeks from the end of radiation therapy performed for clinical or radiological (RECIST 1.1) disease persistence/progression/recurrence with tumour present/unknown on final pathology.
Response Rate evaluated by RECIST | 6 years
Number and Severity of Adverse Events | 6 years
Patient Reported Outcomes utilizing PRO-CTCAE | 6 years
  We will qualitatively compare PRO-CTCAE item scores between arms at 8 weeks from the start of RT, and examine PRO-CTCAE item scores at 12 months post-RT in the SBRT arm, as an indicator or persisting (consequential or "late") RT toxicity with SBRT to the head and neck region.
Patient Reported Outcomes utilizing FACT-HN | 6 years
  proportion of patients between arms who have a meaningful worsening (12 points or greater) of QOL
Healthcare Resource Utilization utilizing EQ-5D-5L | 6 years
  All enrolled participants who have received at least one fraction of protocol therapy are evaluable for health economics. Those who have completed the Health Utilities Index (EQ-5D-5L), will be evaluable for cost-utility analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Poon, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences, UHN, Toronto, ON Canada
Locations (5):
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG Policy
URL: https://www.ctg.queensu.ca/public/policies